CLINICAL TRIAL: NCT01491711
Title: Treatment of Superficial Basal Cell Carcinoma by Topical Photodynamic Therapy With Fractionated 5-aminolevulinic Acid 20% Versus Two Stage Topical Photodynamic Therapy With Methylaminolevulinate
Brief Title: Superficial Basal Cell Carcinoma Treatment With Topical Photodynamic Therapy With Fractionated 5-aminolevulinic Acid 20% Versus Two Stage Methylaminolevulinate
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other); VieCuri Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL38127
Record Dates: First submitted 2011-12-05; First posted 2011-12-14 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Superficial Basal Cell Carcinoma
Keywords: Superficial basal cell carcinoma; Carcinoma, Basal Cell; Skin diseases; Connective tissue diseases; Treatment; Drug therapy; Efficacy; Photodynamic therapy; Photosensitizing Agents/therapeutic use; Aminolevulinic acid; Methylaminolevulinate; Pain measurement; Health Care Economics and Organizations
MeSH Terms: conditions — Carcinoma, Basal Cell; Skin Diseases; Connective Tissue Diseases | interventions — methyl 5-aminolevulinate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fractionated 5-ALA HCl 20% gel PDT (Active Comparator): Twice on day 1
  Interventions: Drug: Fractionated 5-aminolevulinic acid hydrochloride 20% gel PDT
- Methylaminolevulinate PDT in 2 sessions (Active Comparator): On day 1 and 8
  Interventions: Drug: Methylaminolevulinate PDT in 2 sessions

INTERVENTIONS:
Drug: Methylaminolevulinate PDT in 2 sessions — The methylaminolevulinate creme is applied to the tumour with a margin of 1 cm, ± 1-2 mm thick. Tegaderm®, a gauze and tinfoil is placed over the area to prevent contact with UV light. After 4 hours the area is illuminated with Aktilite (632 nm, 570-670 nm, 75 J/cm2). The light intensity at the lesion surface should not exceed 200 mW/cm2. During illumination a fan is used to cool the treatment site. After the first treatment the skin area is covered to prevent exposure to daylight during 48 hours. After one week (on day 8), the same procedure is repeated. After the treatment the skin area is covered to prevent exposure to daylight during 48 hours. A side-effect of the treatment is a burning pain during illumination and slight erythema afterwards lasting a few days. Sometimes blistering occurs.
  Other Names: Metvix 160 mg/g creme; CAS number 33320-16-0; ATC code L01XD03; RVG 31130
  Arms: Methylaminolevulinate PDT in 2 sessions
Drug: Fractionated 5-aminolevulinic acid hydrochloride 20% gel PDT — The 5-ALA HCl 20% gel is applied to the tumour with a margin of 1 cm, ± 1-2 mm thick. Tegaderm®, a gauze and tinfoil is placed over the area to prevent contact with UV light. After 4 hours the area is illuminated with Aktilite (632 nm). During illumination a fan is used to cool the treatment site. The treatment site is covered again with Tegaderm for 2 hours after first treatment, whereupon a second illumination with the same light takes place. A side-effect of the treatment is a burning pain during illumination and slight erythema afterwards lasting a few days. Sometimes blistering occurs. Patients are advised to avoid direct sunlight two days after treatment.
  Arms: Fractionated 5-ALA HCl 20% gel PDT

SUMMARY:
Skin cancer is the most common cancer in Caucasians, and a basal cell carcinoma (BCC) being the most common skin cancer with around 44,000 new tumours per year, and its incidence is still rising. In the past it has been a disease of the elderly patient but as a consequence of recreational sun exposure and tanning beds, more young patients develop a skin cancer as well. There are different subtypes of BCC and most subtypes are treated by surgical excision. Nowadays, non-invasive techniques as photodynamic therapy (PDT) are common practice to treat superficial BCC (sBCC). Because of these techniques treatment by surgical excision can be avoided with the possibility of complications and scar formation. Both 5-aminolevulino acid (5-ALA) and the more lipophilic methyl aminolevulinate (MAL) can be used as a precursor of the photosensitiser. These agents generate an excess of protoporphyrin IX in metabolic active cells, which are illuminated by a specific light source leading to release of reactive oxygen radicals in tissue. The result is apoptosis and necrosis of tumour cells. At the moment, two treatment protocols are used in the Netherlands: the fractionated 5-ALA 20% (Fagron) protocol according to de Haas and the MAL (Metvix, Galderma) protocol. Because MAL was first marketed and registered as a treatment option for premalignant and superficial malignancies most hospitals in the Netherlands use this topical agent. However, there is no evidence which of the 2 agents is more (cost-)effective and/ or preferred by patients.

Objective: to determine which treatment is the most effective treatment in terms of prevention of treatment failure, cost saving and patients preference when comparing fractionated 5-ALA 20% PDT versus MAL PDT in 2 treatment sessions.

DETAILED DESCRIPTION:
- Basal cell carcinoma throughout the world

Skin cancer is the most common form of cancer, with basal cell carcinoma (BCC) being the most common form of all skin cancers, and the incidence is still rising.1,2 Of all types of BCC, superficial basal cell carcinoma (sBCC), is the histopathologic subtype with the fastest growing incidence, especially on the trunk in younger patients.3-5 It is a common health problem and although there is no chance of metastasis it can lead to more aggressive forms of BCC with the ability to cause serious local destruction.

- Treatment options

The DBC (diagnose behandel combinatie) cost price, the amount received for diagnostic and treatment of one BCC, for surgical excision is partly free negotiable between each hospital and health insurances. Only the DBC cost price of patients whose health insurance has no contract with the hospital is public for everyone. This leads to around 18 million euro (based on a cost price of 400.00 euro for 44,000 new BCCs per year) that is yearly spent on the surgical treatment of BCC in the Netherlands and cost will only increase in future with the growing incidence.6 For most BCC subtypes the only effective treatment is surgery but for sBCC other non-invasive treatments like photodynamic therapy (PDT) are suitable. It is well accepted in today's dermatologic practice that surgical excision can be considered as over-treatment for sBCC.7-9 PDT is superior to surgical excision in primary sBCC of any size in low-risk sites.9 As a consequence unnecessary anaesthesia and incisions are avoided thereby preventing side-effects, such as scars, haematomas or functional disruption, and healthy tissue is preserved. MAL is a worldwide registered agent for the use of topical PDT in sBCC while 5-ALA is not registered in the European Union. In the Netherlands both fractionated 5-ALA 20% and MAL PDT in 2 sessions are used as treatment for sBCC. Although there are studies showing the effectiveness of both treatment regimens, the effectiveness, costs and patient preferences have never been studied in a prospective randomised trial.

- Developments in treatment: photodynamic therapy

PDT has become increasingly implemented in standard care for sBCC in the last years.8-10 Nowadays, in the Maastricht University Medical Centre, about 60% of patients are treated with PDT. Similar situations are found in the Erasmus MC Rotterdam and the VieCuri Medical Centre Venlo/Venray. On national level, around two thirds of patients are treated with MAL PDT in 2 sessions and one third with fractionated 5-ALA 20% PDT. This distribution is historically determined and not based on evidence based research.

- 5-ALA 20% PDT versus MAL PDT

There are only a few randomised controlled studies on treatment of the most common skin cancer.11 Choice of PDT treatment with fractionated 5-ALA 20% or MAL in 2 sessions often depends on the experience and choice of the physician or the availability of the precursor in a hospital. World-wide, most studies are performed with MAL and it has been accepted as the standard of care in PDT.12 However, according to the literature, the effectiveness in terms of clearance rates is in different studies lower for MAL in two sessions compared to fractionated 5-ALA 20% PDT: 79% versus 97% intention to treat (ITT) after one year in sBCC.13,14 Contra dictionary, MAL has the theoretical benefit of being more and faster absorbed in the cell than 5-ALA 20% and, thereby, should generate a higher production of protoporphyrin IX. In addition MAL has higher selectivity for tumour cells, inducing fewer side-effects in normal tissue. 15,16 This discrepancy between theoretical working mechanism and clearance rates needs further clinical research of the effectiveness of both treatments.

PDT is a hospital administered treatment modality during which patients have to come to the hospital one day (fractionated 5-ALA 20%) or two days one week apart (MAL in 2 sessions). Patient compliance could be higher with fractionated 5-ALA 20% than with MAL in 2 sessions because patients have to visit the hospital a second time. At some parts of the body patients experience a variable burning pain sensation during PDT which might influence completing the treatment. Kuijpers et al. found no significant differences in pain scores between ALA-PDT in 2 sessions and MAL PDT in 2 sessions.17 We expect 5-ALA 20% PDT to have more side-effects in our study as patients are treated twice on the same day.

Furthermore it is important to take into consideration the differences in patient acceptability costs (see 'economic evaluation').18 A well-designed study comparing the two topical PDT treatment modalities: fractionated 5-ALA 20% and MAL in 2 sessions will provide the answers needed to establish the position of the two modalities in the treatment of patients with sBCC. The conclusions from the proposed study can serve as a basis for updating guidelines for the treatment of sBCC to catch up with recent developments in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Minimal age of 18 years
* Histological proven BCC
* Primary BCC (no previous treatment)
* Being able to understand instructions

Exclusion Criteria:

* Age under 18 years
* No histological proven BCC
* Recurrent BCC (previously treated)
* Not able to understand instructions
* Concomitant disease requiring systematic immunosuppressive treatment
* Genetic skin cancer disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | 12 months posttreatment
  Histological proven treatment failure one year after treatment of sBCC with fractionated 5-ALA 20% PDT versus MAL PDT in 2 sessions. If there is any clinical suspicion of residual tumour at control visits 3 and 12 months posttreatment, a 3 mm punch biopsy will be taken to confirm the diagnosis by histopathology.

SECONDARY OUTCOMES:
Patient preferences | 1 week posttreatment
  Patient preferences of treatment with fractionated 5-ALA 20% PDT versus MAL PDT in 2 sessions.
  A patient questionnaire will be given twice: on last day of treatment and 1 week posttreatment
Health care costs | 12 months posttreatment
  Health care costs of treatment with fractionated 5-ALA 20% PDT versus MAL PDT in 2 sessions.

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Maastricht University Medical Center, Maastricht, Limburg
  - VieCuri Medical Centre, Venlo, Limburg
  - Erasmus Medical Centre, Rotterdam, South Holland